CLINICAL TRIAL: NCT00894504
Title: A Phase II Trial of Panitumumab, Gemcitabine, and Carboplatin in Triple-Negative Metastatic Breast Cancer
Brief Title: Panitumumab, Gemcitabine and Carboplatin in Triple-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Amgen (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 126
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic Breast Cancer; Triple Negative; Panitumumab; Vectibix; Gemcitabine; Gemzar; Carboplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — Panitumumab; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab/Gemcitabine/Carboplatin (Experimental): Systemic therapy
  Interventions: Drug: Panitumumab; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Panitumumab — 6 mg/kg IV on Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks)
  Other Names: Systemic Therapy; Vectibix
Drug: Carboplatin — AUC=2.5 IV, Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks)
  Other Names: Systemic Therapy; Paraplatin
Drug: Gemcitabine — 1500 mg/m2 IV, Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks)
  Other Names: Systemic Therapy; Gemzar

SUMMARY:
In this Phase II trial, the investigators will evaluate the combination of gemcitabine, carboplatin, and panitumumab in the treatment of patients with metastatic triple-negative breast cancer. In addition, to assess the efficacy of this combination, tumor tissue will be examined for the presence of various markers, including K-ras and PI3K-activating mutations, EGFR, PTEN, and p53. Correlation of tumor response with marker expression may define a patient subset that is particularly responsive to treatment with a panitumumab-containing combination.

DETAILED DESCRIPTION:
All patients will receive a pre-emptive skin care regimen during panitumumab therapy to reduce skin toxicity. Treatment cycles will be repeated every 14 days (2 weeks). During each treatment, panitumumab will be administered first, then carboplatin, then gemcitabine. All drugs will be administered according to standard guidelines. Patients will be re-evaluated for response after completion of 3 cycles (6 weeks) of treatment. Patients with objective response or stable disease will continue treatment. Subsequent re-evaluations will occur every 6 weeks. Patients will continue treatment with all three drugs until tumor progression, or until unacceptable toxicity occurs. If patients experience toxicity caused by gemcitabine/carboplatin and are continuing to benefit from treatment, panitumumab can be continued as a single agent (at the same dose and schedule), at the discretion of the investigator, until disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients >=18 years of age.
2. Histologically or cytologically confirmed diagnosis of unresectable locally advanced or stage IV breast cancer.
3. No more than 1 prior treatment regimen for metastatic breast cancer.
4. Estrogen receptor and progesterone receptor negative (defined as <10% staining by IHC).
5. Paraffin-embedded tumor tissue (from the primary tumor or metastasis) for biomarker testing. (In the absence of paraffinembedded tissue, unstained paraffin-embedded tumor slides are acceptable).
6. Measurable disease, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) guidelines
7. HER2 negative tumors. HER2 negativity must be confirmed by one of the following:

   * FISH-negative (FISH ratio <2.2), or
   * IHC 0-1+, or
   * IHC 2-3+ AND FISH-negative (FISH ratio <2.2)
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1.
9. Absolute neutrophil count (ANC) >=1.5 × 109/L; platelet count >=100 × 109/L; hemoglobin >=9.0 g/dL.
10. Creatinine <=1.5 mg/dL, or creatinine clearance >=40 mL/min (as calculated by the Cockcroft-Gault method, as follows: Female creatinine clearance = (140 - age) × (weight in kg) × 0.85 (serum creatinine × 72)
11. Adequate hepatic function, defined as follows: total bilirubin <=1.5 x ULN; aspartate aminotransferase (AST) <=3 × ULN (or <= 5 x ULN if liver metastases); alanine aminotransferase (ALT) <=3 x ULN (or <=5 x ULN if liver metastases).
12. Magnesium level >= the institutional lower limit of normal (LLN).
13. Women of childbearing potential must agree to use adequate contraception (per institutional standard of care) during treatment and until 6 months after the last administration of investigational products.

Exclusion Criteria:

1. Patients with brain metastases are not eligible.
2. History of another primary cancer, with the exception of the following:

   * Curatively treated in situ cervical cancer;
   * Curatively resected non-melanoma skin cancer;
   * Other primary solid tumor curatively treated with no known active disease present and no treatment administered for >=5 years prior to study enrollment.
3. History of interstitial lung disease (e.g., pneumonitis, pulmonary fibrosis), or any evidence of interstitial lung disease on the CT scan of the chest performed at the baseline visit.
4. Prior anti-EGFR antibody therapy (e.g., cetuximab), or treatment with small-molecule EGFR inhibitors (e.g., gefitinib, erlotinib, lapatinib).
5. Radiotherapy <=14 days prior to study enrollment. Any acute effects of radiotherapy must be resolved prior to the administration of study drugs.
6. Systemic chemotherapy, hormonal therapy, immunotherapy, or experimental or approved proteins/antibodies (e.g., bevacizumab) <=21 days prior to study enrollment.
7. Prior therapy with gemcitabine or carboplatin in the metastatic setting is not permitted. Patients who received gemcitabine or carboplatin as part of adjuvant therapy are eligible, as long as recurrence was first documented >12 months after the last exposure to the drug(s).
8. Major surgery within 28 days or minor surgery within 14 days of study enrollment.
9. Requirement of chronic use of immunosuppressive agents (e.g., methotrexate, cyclosporine).
10. Any investigational agent or therapy <=30 days prior to study enrollment.
11. Uncontrolled or intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
12. History of any medical or psychiatric condition or laboratory abnormality that, in the opinion of the investigator, may increase the risks associated with the study participation or administration of the investigational products, or that may interfere with the interpretation of the results.
13. Unwillingness or inability to comply with study requirements.
14. Women who are pregnant or breastfeeding.
15. Patients with known human immunodeficiency virus (HIV), hepatitis C virus, and/or acute or chronic hepatitis B virus infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2010-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise A Yardley, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (17):
- United States (17):
  - Los Robles, Thousand Oaks, California
  - Aventura Hospital and Medical Center, Aventura, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Nebraska Methodist Cancer Center, Omaha, Nebraska
  - Atlantic Health System, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Health Physician Group, Dallas, Texas
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Panitumumab/Gemcitabine/Carboplatin: Treatment cycles are repeated every 14 days (2 weeks)
  Panitumumab: 6mg/kg intravenous (IV), Day 1 of each 2-week treatment cycle.
  Gemcitabine: 1500mg/m2 IV, Day 1 of each 2-week treatment cycle
  Carboplatin: Area Under the Curve (AUC) = 2.5 IV, Day 1 of each 2-week treatment cycle
Period: Overall Study
Arm/Group | Panitumumab/Gemcitabine/Carboplatin
Started | 71
Completed | 0
Not Completed | 71

BASELINE CHARACTERISTICS:
Groups:
- Panitumumab/Gemcitabine/Carboplatin: Panitumumab - 6 mg/kg IV on Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks) Carboplatin - AUC=2.5 IV, Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks) Gemcitabine - 1500 mg/m2 IV, Day 1 of each 2-week treatment cycle for 3 cycles (6 weeks)
Arm/Group | Panitumumab/Gemcitabine/Carboplatin
Number analyzed (Participants) | 71
Age, Continuous [Median (Full Range); unit: Years] | 54 [32 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Measured from Day 1 of study drug administration to disease progression - defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 as a 20% increase in the sum of the longest diameter of target lesions and/or appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions
Time Frame: every 6 weeks until treatment discontinuation
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Panitumumab/Gemcitabine/Carboplatin
Number analyzed (Participants) | 71
Months | 4.4 [3.2 to 5.5]

2. Secondary Outcome: Objective Response Rate and Clinical Benefit Rate
Description: Estimated as the proportion of subjects who meet the criteria for complete or partial response (CR or PR) per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1 - for target lesions assessed by MRI: Complete Response (CR) is defined as disappearance of all target lesions; Partial Response (PR) is defined as >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: every 6 weeks until treatment discontinuation
Population: All evaluable patients per RECIST v 1.1
Measure: Number; unit: Participants
Arm/Group | Panitumumab/Gemcitabine/Carboplatin
Number analyzed (Participants) | 69
Participants
  Clinical benefit rate (CR + PR + SD>6 months) | 32
  Objective response rate (CR + PR) | 30

3. Secondary Outcome: Number of Treatment-related Toxicities Occurring in ≥10% of Patients as a Measure of Tolerability and Toxicity
Description: Assessments made through analysis of treatment-related adverse events and serious adverse events
Time Frame: every 6 weeks until discontinuation of treatment, expected average of 18 months
Measure: Number; unit: participants
Arm/Group | Arm/Group 1
Number analyzed (Participants) | 71
participants
  Neutropenia | 32
  Thrombocytopenia | 32
  Leukopenia | 25
  Anemia | 20
  Rash | 50
  Fatigue | 37
  Nausea/vomiting | 36
  Dry skin | 21
  Hypomagnesemia | 18
  Mucositis/stomatitis | 16
  Constipation | 15
  Dyspnea | 12
  Pruritis | 12
  Anorexia | 10
  Diarrhea | 9
  AST/ALT increased | 9
  Alopecia | 7
  Dyspepsia | 7
  Myalgia | 7

4. Secondary Outcome: Correlation of Biomarker Expressions of EGFR, K-ras, p53, PTEN Expression, and PI3K in Triple-negative Breast Cancer With Response to Treatment With the Combination of Gemcitabine, Carboplatin, and Panitumumab
Description: Median PFS (95% CI), months, reported by biomarker expression/mutation status for: EGFR, p53, PTEN, PIK3CA, KRAS
Time Frame: 18 months
Population: Excludes patients in the following categories due to insufficient data: PTEN status unknown, PIK3CA Status unknown and KRAS no mutation
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EGFR Normal | EGFR Amplified | p53 Normal | p53 Loss | PTEN Normal | PTEN Loss | PIK3CA No Mutation | PIK3CA Mutation(s)
Number analyzed (Participants) | 56 | 12 | 34 | 34 | 62 | 5 | 55 | 12
months | 4.57 [3.88 to 6.44] | 3.42 [1.51 to NA] — Upper limit of 95% Confidence Interval not available - too few patients in this category | 4.16 [2.69 to 5.49] | 5.32 [3.19 to 9.03] | 4.4 [3.88 to 5.59] | 2.91 [0.82 to NA] — Upper limit of 95% Confidence Interval not available - too few patients in this category | 4.37 [3.19 to 6.05] | 4.73 [2.56 to NA] — Upper limit of 95% Confidence Interval not available - too few patients in this category

ADVERSE EVENTS:
Arm/Group | Panitumumab/Gemcitabine/Carboplatin
Serious Adverse Events (participants affected / at risk) | 10/71
Other Adverse Events (participants affected / at risk) | 70/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab/Gemcitabine/Carboplatin (N=71)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
CARDIAC TAMPONADE (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (2)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
CHEST PAIN (General disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (3)
EMBOLISM (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab/Gemcitabine/Carboplatin (N=71)
ANAEMIA (Blood and lymphatic system disorders) | 16 (46)
LEUKOPENIA (Blood and lymphatic system disorders) | 18 (114)
NEUTROPENIA (Blood and lymphatic system disorders) | 24 (121)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 25 (54)
TACHYCARDIA (Cardiac disorders) | 6 (8)
DRY EYE (Eye disorders) | 4 (4)
CONSTIPATION (Gastrointestinal disorders) | 28 (41)
DIARRHOEA (Gastrointestinal disorders) | 13 (26)
DYSPEPSIA (Gastrointestinal disorders) | 7 (9)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 (6)
NAUSEA (Gastrointestinal disorders) | 38 (56)
STOMATITIS (Gastrointestinal disorders) | 7 (8)
VOMITING (Gastrointestinal disorders) | 17 (28)
FATIGUE (General disorders) | 45 (109)
MUCOSAL INFLAMMATION (General disorders) | 9 (22)
OEDEMA PERIPHERAL (General disorders) | 5 (5)
PYREXIA (General disorders) | 7 (8)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 7 (40)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 (32)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (20)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4 (19)
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 (26)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (8)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 (17)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 8 (14)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 16 (29)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 6 (8)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4 (21)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (8)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 (6)
DIZZINESS (Nervous system disorders) | 5 (6)
DYSGEUSIA (Nervous system disorders) | 6 (6)
HEADACHE (Nervous system disorders) | 6 (8)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 8 (10)
ANXIETY (Psychiatric disorders) | 7 (8)
DEPRESSION (Psychiatric disorders) | 4 (4)
INSOMNIA (Psychiatric disorders) | 12 (12)
DYSURIA (Renal and urinary disorders) | 5 (5)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (13)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 14 (21)
ACNE (Skin and subcutaneous tissue disorders) | 6 (11)
ALOPECIA (Skin and subcutaneous tissue disorders) | 7 (7)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 8 (17)
DRY SKIN (Skin and subcutaneous tissue disorders) | 24 (28)
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 6 (13)
PRURITUS (Skin and subcutaneous tissue disorders) | 11 (13)
RASH (Skin and subcutaneous tissue disorders) | 31 (55)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites